CLINICAL TRIAL: NCT02626884
Title: Ibrutinib in Relapsed Nodular Lymphocyte-predominant Hodgkin Lymphoma (NLPHL)
Acronym: IRENO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Engert, Prof., University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1776; 2015-003128-30 (EudraCT Number)
Record Dates: First submitted 2015-12-02; First posted 2015-12-10 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Nodular Lymphocyte-Predominant Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibrutinib (Experimental): All patient receive ibrutinib at a dose of 560 mg/d for up to 20 21-day cycles
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib

SUMMARY:
The purpose of this trial is to determine

1. Disease stabilization/response rate after six 21-day cycles of ibrutinib
2. Remission status after six, twelve and 20 21-day cycles of ibrutinib

ELIGIBILITY:
Inclusion Criteria (key criteria):

1. Histologically proven relapsed nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL) as confirmed by expert review
2. Age at entry 18-99 years
3. ECOG status 0-2
4. Absolute leukocyte count > 2.500/mm3
5. Absolute neutrophil count > 1.000/mm3 independent of growth factor support
6. Platelet count > 100.000/mm3 or > 50.000/mm3 in case of bone marrow involvement independent of transfusion support in either situation
7. GPT and GOT ≤ 3 x upper limit of normal (ULN)

Exclusion Criteria (key criteria):

1. Classical HL (cHL) or composite lymphoma
2. Known central nervous lymphoma
3. Prior Btk inhibitor treatment
4. Life expectancy < 3 months
5. Major surgery within 4 weeks of study inclusion
6. History of stroke or intracranial hemorrhage within 6 months prior to the first study drug
7. Current anticoagulation with warfarin or equivalent vitamin K antagonists

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Response Rate | after 6 cycles (each cycle is 21 days) of Ibrutinib

SECONDARY OUTCOMES:
Remission status | Remission status after six, twelve and 20 21-day cycles of ibrutinib

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — University Hospital of Cologne
Locations (1):
- 1st Department of Medicine, Cologne University Hospital, Cologne, Germany